CLINICAL TRIAL: NCT01650350
Title: Low Dose Naltrexone for Metastatic Melanoma, Castrate Resistant Prostate Cancer and Renal Cancer: A Phase II Brown University Oncology Group Research Project
Brief Title: Low Dose Naltrexone for Metastatic Melanoma, Castrate Resistant Prostate Cancer and Renal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped 10/24/13 secondary to lack of patients/slow enrollment
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 275
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Melanoma; Prostate Cancer; Renal Cancer
Keywords: Melanoma; Prostate Cancer; Renal Cancer
MeSH Terms: conditions — Melanoma; Prostatic Neoplasms; Kidney Neoplasms | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low Dose Naltrexone (Experimental): LDN, 5 mg/day-(1 cycle = 28 days).
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — 4.1 Low Dose Naltrexone (LDN) LDN, 5 mg/day, at approximately 9pm, on an empty stomach, until disease progression, unacceptable toxicity, need for initiation of narcotic analgesia, or removal from protocol treatment according to section 12.0. (1 cycle = 28 days).
  LDN, 5mg/ml, will be prepared by the Lifespan hospital pharmacy for patient use for this study.
  Other Names: Revia and Vivitrol

SUMMARY:
will scientifically evaluate whether Low Dose Naltrexone (LDN) has activity in refractory solid tumors within the context of a phase II clinical study

DETAILED DESCRIPTION:
Three types of solid tumors will be studied in this protocol: Melanoma, castrate resistant prostate cancer and kidney cancer. Systemic chemotherapy may weaken the immune system reducing the potential for response to LDN. Therefore, patients must either have not had previous chemotherapy or patients must not have received more than 1 prior chemotherapy regimen which must have been completed at least 6 months prior to LDN. Systemic chemotherapy has at best modest activity in melanoma, CRPC and renal cancer.

* Melanoma will be evaluated since the responding patient at the Miriam Hospital had melanoma. Immunomodulatory agents such as ipilimumab have already demonstrated a survival advantage in melanoma.
* Castrate Resistant Prostate Cancer (CRPC): It is common in CRPC for patients to have rising PSA after failure of androgen deprivation. These patients may be asymptomatic or minimally symptomatic and there is reluctance to initiate treatment with systemic chemotherapy with standard docetaxel since this agent has substantial toxicity and will impair quality of life. Waiting until symptomatic disease progression in patients with CRPC and rising PSA is a commonly utilized strategy. These patients are excellent candidates for a treatment with minimal toxicity such as LDA. The immunomodulatory agent Sipuleucel also improves survival in prostate cancer suggesting that an agent such as LDN could also be helpful.
* Renal cancer will also be studied since this is a disease that has activity with immunomodulants such as IL-2 and interferon. Targeted therapies are generally used for renal cancer. Chemotherapy has minimal activity so most patients are chemotherapy-naive.

ELIGIBILITY:
Conditions for Patient Eligibility

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Histologically or pathologically confirmed melanoma, renal cancer or prostate cancer.
* Patients with melanoma or renal cancer must have metastatic disease.
* Patients with melanoma or renal cancer must have radiographically measurable advanced disease. Patients with measurable cutaneous lesions are also evaluable patients with prostate cancer must be castrate refractory and must have radiographically assessable metastatic disease or must have rising PSA on two sequential measurements.
* No prior chemotherapy, or have not received cytotoxic chemotherapy within the 6 months prior to entry..
* No radiation for 3 weeks prior to beginning Naltrexone
* No requirement for opioid analgesics orNo use of opioid analgesics for at least 10 days.
* Absolute neutrophil count ≥ 1,000/uL, platelet ≥ 75,000/uL.
* Total bilirubin ≤ 1.5x upper institutional limit (ULN) and AST or ALT ≤ 3x ULN;
* No prior history of hepatic failure, cirrhosis or hepatic encephalopathy
* ECOG performance status 0 to 2.
* Creatinine < 1.5 x ULN
* Life expectancy of at least 8 weeks.
* Age ≥ 18 years
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 1 months thereafter.
* Voluntary written informed consent.
* Conditions for Patient Ineligibility Patients meeting any of the following exclusion criteria are not to be enrolled in the study.
* Must not have uncontrolled severe, intercurrent illness.
* Women who are breast-feeding.
* Patients who have undergone major surgery or radiotherapy within the last 3 weeks.
* Patients on concurrent anticancer therapy.
* Patients with known, untreated brain metastasis
* Co-medication that may interfere with study results; e.g opioids
* Known hypersensitivity to any component of naltrexone
* Current or prior alcohol dependence
* Patients who could benefit from conventional therapy are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Director — Brown University
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Naltrexone: LDN, 5 mg/day-(1 cycle = 28 days).
  Naltrexone
Period: Overall Study
Arm/Group | Low Dose Naltrexone
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Dose Naltrexone
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 79.4 [68 to 89]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Responses to Low Dose Naltrexone for Patients With Advanced Melanoma, Castrate Refractory Prostate Cancer (CRPC) or Renal Cancer Via RECIST
Description: Response will be assessed via RECIST 1.1 criteria utilizing interval CT scans and physical exam after every 3 cycles of treatment (i.e. every 12 weeks).
Time Frame: approximately every 3 months CT, every month physical, up to 6 months
Measure: Number; unit: participants
Groups:
- Melanoma: Low Dose Naltrexone; Prostate Cancer- Low Dose Naltrexone: LDN, 5 mg/day-(1 cycle = 28 days).
  Naltrexone
Arm/Group | Melanoma: Low Dose Naltrexone | Prostate Cancer- Low Dose Naltrexone
Number analyzed (Participants) | 1 | 6
participants
  stable disease by RECIST | 0 | 2
  progression of disease by PSA | 0 | 6
  progression via RECIST | 0 | 1
  progression clinical | 1 | 0

2. Secondary Outcome: To Assess the Toxicity Associated With Low Dose Naltrexone for Melanoma, CRPC and Renal Cancer.
Description: Defined by number of patients who experienced a SAE
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Naltrexone
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: Monthly and 30 days post last dose of drug (approximately 9 months)
Arm/Group | Low Dose Naltrexone
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Naltrexone (N=7)
Anemia (Investigations) | 4 (4)
RBC (Investigations) | 1 (1)
infection (Investigations) | 1 (1)
abd pain (Investigations) | 1 (1)
kidney pain (Investigations) | 1 (1)
fatigue (Investigations) | 3 (3)
anorexia (Investigations) | 2 (2)
nausea (Investigations) | 1 (1)
upset stomach (Investigations) | 1 (1)
diarrhea (Investigations) | 1 (1)
leg cyst (Investigations) | 1 (1)
LFT (Investigations) | 1 (1)
seg neutrophils (Investigations) | 1 (1)
constipation (Investigations) | 1 (1)
dyspnea (Investigations) | 1 (1)
achilles pain (Investigations) | 1 (1)
pain scalp (Investigations) | 1 (1)
scalp lesion- Moh's (Investigations) | 1 (1)
weight loss (Investigations) | 1 (1)
PLT (Investigations) | 1 (1)
Rash- thigh (Investigations) | 1 (1)
creatinine (Investigations) | 1 (1)
edema (Investigations) | 1 (1)
Pain- shoulder (Investigations) | 1 (1)
pain-hip (Investigations) | 1 (1)
insomnia (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No